CLINICAL TRIAL: NCT03713385
Title: Comparison Between the Subglotic Diameter and the Epiphyseal Diameter of the Radius in Children for Prediction of Appropriate Endotracheal Tube Sizes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nevert Adel, lecturer of anesthesia, surgical ICU and pain management, Mansoura University
Other Study IDs: MansouraU4
Record Dates: First submitted 2018-10-18; First posted 2018-10-19 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Prediction of Pediatric Endotracheal Tube Size

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aged group (n =49): Determined the optimal endotracheal tube size according to age of the child (internal diameter [ID] in mm = [age in years + 16] /4) suggested by Cole
- Subglottic diameter group (n =49): The subglottic transverse diameter was estimated with ultrasonography on the middle of the anterior region of the neck at the level of cricoid cartilage
- Epiphyseal diameter group (n =49): The epiphyseal transverse diameter of the distal radius was estimated with ultrasonography.

SUMMARY:
Background: In pediatric anesthesia, selection of the appropriate endotracheal tube (ETT) size is an important task because the inappropriate one may lead to much complication. The aim of this study is to compare between the subglotic diameter and the epiphysis diameter of radius measured by ultrasonography for prediction of optimum endotracheal tube size in children.

Methods: Patients aged from 1 to 6 years will be scheduled for elective surgery under general anesthesia and intubation, were enrolled in this study. Patients were randomly divided into three groups according to method of choosing the tube size.

Aged group (n =49): determined the optimal endotracheal tube size according to age of the child (internal diameter [ID] in mm = [age in years + 16] /4) suggested by Cole.4 Subglottic diameter group (n =49): The subglottic transverse diameter was estimated with ultrasonography on the middle of the anterior region of the neck at the level of cricoid cartilage.

Epiphyseal diameter group (n =49): the epiphyseal transverse diameter of the distal radius was estimated with ultrasonography.

Patient descriptive data, size of the selected ETT, number and size of the optimum tube, number of re-intubation due to incorrect size of ETT either smaller or larger were recorded. Subglottic transverse diameter (mm) and time of intubation were measured. After intubation, pulse, respiratory rate, arterial blood saturation, capnograghy and airway pressure were recorded during surgery.

Any airway complications after extubation as edema, stenosis or stridor were also recorded.

DETAILED DESCRIPTION:
Introduction:

In pediatric anesthesia, selection of the appropriate endotracheal tube (ETT) size is an important task because the inappropriate one may lead to much complication. Oversized tubes cause airway edema, post- extubation stridor, subglottic stenosis, or cartilaginous ischemia, smaller ones increase the resistance to gas flow and risk of aspiration, insufficient ventilation, and poor monitoring of end tidal gases.Therefore, many methods have been suggested recently to precisely predict the optimal size of ETT in children to avoid any harmful complication.

Most of the anesthesiologists choose the appropriate ETT size by using calculating formulae which are based on the children's descriptive data such as weight, height or age. The Cole's equation (internal diameter [ID] in mm = [age in years + 16] / 4) is still considered as one of the prevalent methods in spite of its poor prediction power.

Bone and cartilage growth of the body are supposed to be related to each other, therefore some measurements of body growth as bony cartilage growth of the hand are worthy of attention as a marker of tracheal diameter specially bone measurements for the hand is generally accepted as the indicator of growth.

Also, the transverse diameter or width of the child's fifth fingernail has been used to select the size of ETT. However, a few reports have stated that it is unreliable method to predict the correct tube.

The epiphyseal transverse diameter of the distal radius measured by ultrasonography is a good predictor of the appropriate ETT size. This formula can be rephrased in a tidy way as follows: ETT (mm) = (29.5 + EpiRad [mm])/8.

The ultrasonography could be a reliable, safe, and non-invasive modality for evaluation of the upper airway at the level of subglottic region which considered the narrowest diameter of upper airway and may be helpful to estimate the proper size endotracheal tube. Ultrasound offers a number of advantages compared to other competitive imaging modalities.

Our proposal:

Is to find the best, easier way and most safe method to select the optimum ETT size for children.

Aim of the work:

To compare between the subglotic diameter and the epiphysis diameter of radius measured by ultrasonography for prediction of optimum endotracheal tube size in children.

Research Gap:

To our knowledge, it is the first study conducted in Egypt to evaluate the value of ultrasonography in selecting the appropriate endotracheal tube size in children.

Hypothesis:

Selecting the ideal endotracheal tube size is a challenging issue needing more appropriate method for selection. Up till now, no ideal method is present and most physicians depend upon roughly calculated formulas for choosing the size. These methods depend mainly upon patients' age. Here, we used ultrasonography as a simple and accurate method.

Patient & Methods:

This study will be done at Mansoura University Children's Hospital over a three month duration starting from October 2018 till January 2019. Informed consents will be obtained from patients' guardians or parents and the participant data will be kept confidential. All participants are free not to participate in the research at any time without penalty.

Sample size:

Sample size was calculated using Medcalc 15.8 (https://www.medcalc.org/). The primary outcome of interest is the incidence of appropriate tube selection. Previous studies found that the incidence of appropriate tube selections were 74.7% using subglottic US, 45.3% for Cole's formula and 90% for epiphyseal diameter (Gnanaprakasam & Selvaraj, 2017; Rajanalini & Anitha, 2018). Using the difference between subglottic & cole's (29.4%): sample size = 49 per group.

Patients aged from 1 to 6 years will be scheduled for elective surgery under general anesthesia and intubation, were enrolled in this study. Patients were randomly divided into three groups (49 patients each) according to method of choosing the tube size.

Aged group (n =49): determined the optimal endotracheal tube size according to age of the child (internal diameter [ID] in mm = [age in years + 16] /4) suggested by Cole.4 Subglottic diameter group (n =49): The subglottic transverse diameter was estimated with ultrasonography on the middle of the anterior region of the neck at the level of cricoid cartilage.

Epiphyseal diameter group (n =49): the epiphyseal transverse diameter of the distal radius was estimated with ultrasonography.

Study design:

A cross sectional observational study.

Technique:

An intravenous cannula was inserted and secured. General anesthesia was induced by inhalation of sevoflurane or intravenous administration of intravenous anesthetic as thiopental sodium (5 mg/kg). Muscular relaxation was achieved with atracurium (0.5mg/kg) to facilitate ETT intubation under direct laryngoscopy. The lungs were ventilated with 100% oxygen via a facemask before intubation.

Size of the initial tube was selected as follows: Aged group determined ETT size according to age of the child (internal diameter [ID] in mm = [age in years + 16]/4) suggested by Cole.4 In subglottic diameter group, the subglottic diameter was estimated with B-mode ultrasonography (Korean, Siemens, Acuson, x300) with a 10-13-MHz linear probe positioned on the midline of the anterior neck. The evaluation began by identifying the true vocal folds as paired hyperechoic linear structures that moved with respiration and swallowing before patients were paralyzed. The probe was then moved caudally to visualize the cricoid arch which appears as an arched, rounded and hypoechoic structure. The transverse air-column diameter was measured at the lower edge of the cricoid cartilage after patients were paralyzed.

The measurements of the subglottic diameter was used to select the size of the outer diameter of ETT by the equation [ETT OD=0.55*(subglottic diameter) +1.16, R2= 0.90 for un-cuffed].9 In epiphyseal diameter group , The epiphyseal transverse diameter of the distal radius was measured by B-mode ultrasonography (Korean, Siemens, Acuson, x300) with a 10-13-MHz linear probe, the internal diameter of ETT was selected by using the equation internal diameter of ETT (mm) = (29.5 + EpiRad [mm])/8 (EpiRad: transverse diameter of the distal radius).

All tracheas were intubated with an uncuffed Mallinckrodt ETT with a Murphy's eye. The tracheal tube place was confirmed by auscultation.

The correct ETT size was considered optimal when an audible air leak around the tube at an inspiratory airway pressure was detected between 10-30 cmH2O, with the head and neck in a neutral position. The presence of an air leak was assessed by closing off the pop-off valve and allowing pressure to rise slowly until an audible leak was heard using a stethoscope. If there was no audible leak when the lung were inflated to a pressure of 30 cm H2O, the tube was exchanged with one that was 0.5 mm smaller. But if a leak occurred at an inflation pressure of less than ten cm H2O, the ETT was exchanged for one with the 0.5 mm larger tube.

Patient descriptive data, size of the selected ETT, number and size of the optimum tube, number of re-intubation due to incorrect size of ETT either smaller or larger were recorded. Subglottic transverse diameter (mm) and time of intubation were measured. After intubation, pulse, respiratory rate, arterial blood saturation, capnograghy and airway pressure were recorded during surgery.

Any airway complications after extubation as edema, stenosis or stridor were also recorded.

Statistical analysis:

All the data from the three groups will be tabulated and compared with each other using the appropriate statistical methods according to the type of values whether parametric or non-parametric. P value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 1 to 6 years
* scheduled for elective surgery under general anesthesia and intubation

Exclusion Criteria:

* Patients refusal
* An anticipated difficult airway,
* Any respiratory disease that might cause airway narrowing
* Pre-exiting laryngeal or tracheal pathology
* Any lesion that could cause airway deformity due to fibrosis or the presence of a neck anatomical pathologies that could affect the ultrasound evaluation of the airway
* Any abnormality in the wrist and radius bone
* Any disease after epiphyseal diameter as Rickets or skeletal dysplasia
* Prolonged surgery more than 90 minutes

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients aged from 1 to 6 years will be scheduled for elective surgery under general anesthesia and intubation in Pediatric Hospital Mansoura University.
Sampling Method: Probability Sample
Enrollment: 147 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
number of the optimum tube size | 3 months
  number of the optimum tube size used in pediatric patients in each group

SECONDARY OUTCOMES:
number of re-intubation | 3 months
  number of re-intubation due to incorrect size of ETT either smaller or larger in each group

OTHER OUTCOMES:
time of intubation | 3 months
  time was taken for intubation in each group
airway complications | 3 months
  airway complications after extubation as edema, stenosis or stridor

CONTACTS AND LOCATIONS:
Locations (1):
- Gamal Zakaria, Al Mansurah, Egypt